CLINICAL TRIAL: NCT04451668
Title: Open Label Study of Safety/Tolerability of Once Nightly FT218 for the Treatment of Excessive Daytime Sleepiness and Cataplexy in Narcolepsy Patients That Have and Have Not Been Previously Maintained on Twice-nightly Sodium Oxybate IR
Brief Title: An Open Label Study of FT218 in Subjects With Narcolepsy
Acronym: RESTORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avadel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLFT218-1901
Record Dates: First submitted 2020-06-23; First posted 2020-06-30 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Narcolepsy; Cataplexy; Excessive Daytime Somnolence; Sleep Disorder; Sleep Disturbance; Sleep Wake Disorders
MeSH Terms: conditions — Narcolepsy; Cataplexy; Disorders of Excessive Somnolence; Sleep Wake Disorders; Parasomnias

STUDY DESIGN:
Intervention Model Description: Open label treatment with FT218 (once nightly sodium oxybate extended release)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FT218 (Experimental): once nightly sodium oxybate extended release oral solution (FT218)
  Interventions: Drug: FT218

INTERVENTIONS:
Drug: FT218 — once nightly sodium oxybate extended release

SUMMARY:
An Open Label Study to Evaluate Long-Term Safety and Tolerability of a Once Nightly Formulation of Sodium Oxybate for Extended-Release Oral Suspension (FT218) and the ability to switch from twice-nightly immediate release sodium oxybate to once-nightly FT218 for the Treatment of Excessive Daytime Sleepiness and Cataplexy in Subjects with Narcolepsy

DETAILED DESCRIPTION:
This study will enroll subjects with narcolepsy, either NT1 or NT2, who completed the FT218 Phase 3 REST-ON study or eligible subjects with narcolepsy currently receiving a stable dose of twice nightly sodium oxybate IR or mixed salts oxybate (regardless of whether they participated in the REST-ON study), or subjects who are naïve to oxybate therapy (i.e., FT218, twice nightly sodium oxybate IR or mixed salts oxybate). Following a screening period, subjects who meet the entry criteria will be enrolled into the study. Subjects who completed the FT218 Phase 3 REST-ON study will initiate treatment with FT218 at 4.5 g and will follow a titration schedule up to the highest tolerate dose (up to 9 g), or the dose deemed effective by the investigator. Subjects previously maintained on twice nightly sodium oxybate IR will initiate FT218 treatment at a dose equivalent or closest to the total gram dose of twice-nightly sodium oxybate IR and then titrate up or down, in accord with safety and effectiveness as determined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Subjects receiving a stable doses of twice-nightly sodium oxybate IR or mixed salts oxybate for at least 4 weeks and are willing to switch to FT218
* Subjects who completed the CLFT218-1501 REST-ON Study in a compliant manner and for whom the Investigator determines would receive benefit from treatment with FT218 and have not started treatment with twice nightly sodium oxybate IR or mixed salts oxybate
* Are treatment naïve to any oxybate therapy (i.e. FT218, twice nightly sodium oxybate IR or mixed salts oxybate)
* Subjects have a diagnosis of narcolepsy, either confirmed prior to the REST-ON study or as confirmed by the Investigator as defined by the International Classification of Sleep Disorders 3 criteria (AASM 2014)
* Willing and able to give written informed consent for study participation. Young adults (16 and 17 years old) who have not reached the age of majority must be capable of giving assent in addition to consent from a legally authorized guardian, as required by local laws and regulations.

Exclusion Criteria:

* Subjects that terminated the CLFT218-1501 REST-ON Study prior to completing Visit 8
* Any use of the following medications during the study: Anticonvulsants, Clonidine, Hypnotics, Anxiolytics, Sedating antihistamines, Antipsychotics, Other experimental medications designed to treat narcolepsy, cataplexy or any other condition, or other medications with significant sedating effects/CNS depressant effects are prohibited for REST-ON and naive patients. Patients on twice nightly sodium oxybate IR on medications in classes listed above may be eligible for enrollment if the subject has been on a stable dose of the prohibited medication in combination with a stable dose of twice nightly sodium oxybate or mixed salts oxybate for at least three months and has demonstrated no AEs, intolerance, or interactions AND is approved to participate by the Medical Monitor. Sedative hypnotics are prohibited regardless.)
* A diagnosis of sleep apnea where AHI is ≥15 and/or current use of CPAP or other devices for sleep apnea.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | 24 months
  Assess the long-term safety and tolerability of FT218 by the number of participants experiencing treatment-related adverse events
Incidence of clinically significant changes in vital signs | 24 months
  Assess the long-term safety and tolerability of FT218 by the number of participants experiencing clinically significant changes in vital signs
Incidence of clinically significant changes in laboratory test results | 24 months
  Assess the long-term safety and tolerability of FT218 by the number of participants experiencing clinically significant changes in laboratory test results

CONTACTS AND LOCATIONS:
Locations (29):
- United States (27):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Stanford Sleep Medicine, Redwood City, California
  - SDS Clinical Trials, Santa Ana, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Delta Waves, Inc., Colorado Springs, Colorado
  - Pulmonary Disease Specialists, PA, Kissimmee, Florida
  - Sleep Medicine Specialists of South Florida, Miami, Florida
  - FL Pediatric Research Institute, Winter Park, Florida
  - NeuroTrials Research Inc, Atlanta, Georgia
  - SleepCare Research Institute, Inc. d/b/a Clinical Research Institute, Stockbridge, Georgia
  - Fort Wayne Neurological, Fort Wayne, Indiana
  - Helene A. Emsellem, MD PC, Chevy Chase, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - St. Luke's Hospital - Sleep Medicine and Research Center, Chesterfield, Missouri
  - Montefiore Sleep-Wake Disorders Center, The Bronx, New York
  - Advanced Respiratory and Sleep Medicine, Huntersville, North Carolina
  - Sleep Management Institute Intrepid Research, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Brian Abaluck Sleep Medicine, Malvern, Pennsylvania
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
  - Comprehensive Sleep Medicine Associates, Sugar Land, Texas
  - Northwest Houston Neurology, Tomball, Texas
  - TPMG Clinical Research Williamsburg, Williamsburg, Virginia
- Canada (2):
  - West Perry Sound Health Center, Parry Sound, Ontario
  - Jodha Tishon Inc., Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roy A, Stern T, Harsh J, Hudson JD, Ajayi AO, Corser BC, Mignot E, Santamaria A, Morse AM, Abaluck B, Ibrahim S, Schweitzer PK, Lancaster K, Dubow J, Gudeman J. RESTORE: Once-nightly oxybate dosing preference and nocturnal experience with twice-nightly oxybates. Sleep Med X. 2024 Aug 15;8:100122. doi: 10.1016/j.sleepx.2024.100122. eCollection 2024 Dec 15. PMID 39263597